CLINICAL TRIAL: NCT01620944
Title: A 48-Week, Randomized, Open-Label Phase 3B Study Comparing the Antiviral Efficacy and Safety of ATV/RTV 3TC With ATV/RTV Plus TDF/FTC In HIV-1-Infected, Treatment-Naïve Subjects, Followed By a 48-Week Period on ATV/RTV Plus 3TC
Brief Title: Open-Label Study Comparing Efficacy and Safety of ATV/RTV+3TC With ATV/RTV+TDF/FTC in HIV-Infected, Treatment Naïve Subjects, Followed by Treatment With ATV/RTV+3TC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-494; 2011-006187-47 (EudraCT Number)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Results first posted 2021-08-06 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: HIV
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir; Lamivudine; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1: ATV/RTVHS+3TC (Experimental)
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Lamivudine
- Arm2: ATV/RTVHS+TDF/FTC (Active Comparator)
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Tenofovir/Emtricitabine

INTERVENTIONS:
Drug: Atazanavir — Capsule, oral, 300 mg, Once daily (QD), 96 weeks
Drug: Ritonavir — Tablets, oral, 100 mg, QD, 96 Weeks
  Other Names: Ritonavir high sensitivity (RTV HS)
Drug: Lamivudine — Tablet, oral, 300 mg, QD, 96 Weeks
  Arms: Arm1: ATV/RTVHS+3TC
Drug: Tenofovir/Emtricitabine — Tablets, oral, 300/200 mg, QD, 48 Weeks
  Arms: Arm2: ATV/RTVHS+TDF/FTC

SUMMARY:
The primary objective of this study in antiretroviral (ARV)-naïve Human immunodeficiency virus 1 (HIV-1) ribonucleic acid infected subjects is to compare the response rate at Week 48 of a daily regimen of Atazanavir (ATV)/ Ritonavir (RTV)HS 300/100 mg combined with either one additional drug [Lamivudine (3TC) 300 mg daily] or 2 additional drugs [Tenofovir/Emtricitabine(TDF/FTC) 300/200 mg daily].

ELIGIBILITY:
Inclusion Criteria

- Signed Written Informed Consent.

i) Freely given informed consent must be obtained from subjects prior to clinical trial participation, including informed consent for any screening procedures conducted to establish subject eligibility for the trial.

ii) A freely given Pharmacokinetics (PK) sub-study consent form must be obtained from the subset of subjects participating in the intensive PK sub-study.

- Target Population.

i) Treatment-naive HIV-1-infected subjects (< 48 hours of any ARV is allowed).

ii) Subjects who have an HIV-1 Ribonucleic acid (RNA) level ≥ 1000 c/mL at screening.

iii) Subjects who have a Antigenic marker of helper/inducer T lymphocytes (CD4) + cell count > 100 cells/mm3.

- Age and Reproductive Status.

i) Men and women, 18 years of age or older (or minimum age as determined by local regulatory or legal requirements).

ii) Women of childbearing potential (WOCBP) must use highly effective methods of birth control for up to 8 weeks after the last dose of investigational product to minimize the risk of pregnancy. WOCBP must follow instructions for birth control for the entire duration of the study including a minimum of 30 days after dosing has been completed.

iii) Acceptable methods of highly effective birth control include:.

A. Condom with spermicide.

B. Diaphragm and spermicide.

C. Cervical cap and spermicide

- Since acceptable and available methods of contraception vary among different countries, participating women may choose their preferred contraceptive method atazanavir AI424494 BMS-232632 Clinical Protocol Date: 31-01-2012 33 based on physician recommendations. Caution is warranted with co-administration of oral contraceptives (ethinyl estradiol and norethindrone).

i) Women must have a negative serum or urine pregnancy test [minimum sensitivity 25 IU/L or equivalent units of Human chorionic gonadotropin (HCG)] within 24 hours prior to the start of investigational product.

ii) Women must not be breastfeeding.

iii) Sexually active fertile men must use highly effective birth control if their partners are WOCBP.

Exclusion Criteria

- Target Disease Exceptions.

i) Subjects who have an HIV-1 RNA level ≥500,000 c/mL at screening.

ii) Screening HIV genotype showing resistance to any component of the study regimen (ATV, RTV, 3TC, TDF/FTC).

iii) Previously documented HIV-2 infection.

- Medical History and Concurrent Diseases.

i) Acute or chronic hepatitis B virus (HBV) or Acute hepatitis C virus (HCV) co-infection.

- Note Chronic co-infection with hepatitis C is not exclusion criteria. Subjects with acute hepatitis C may have the option to be screened after the event has evolved into a chronic infection.

i) Presence of a newly diagnosed HIV-related opportunistic infection (OI) or any medical condition requiring acute therapy at the time of enrollment. Subjects on stable maintenance therapy for an OI may be enrolled.

ii) Primary HIV infection.

iii) History or current cardiac disease, defined by presence of arrhythmias, ischemic disease, or a conduction abnormality including left bundle branch block (LBB) or left anterior fascicular block (LAFB), 2nd or 3rd-degree atrioventricular block (AVB), or any cardiac abnormality deemed clinically significant by the investigator. In addition, the following Electrocardiogram (ECG) findings are exclusionary:.

A. PR Interval > 260 msec (severe 1st degree AV Block).

B. QRS Interval > 120 msec.

iv) Moderate-to-severe hepatic insufficiency.

v) Obstructive liver disease.

vi) Recent therapy with agents having significant systemic myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic or cytotoxic potential within 3 months of study start or the expected need for such therapy at the time of enrollment, or therapy with methadone or ribavirin/interferons or treatment with neurotoxic drugs or drugs that affect CYP3A4.

vii) Concomitant administration of a proton pump inhibitor (PPI) or H2 blocker or any other drug with potential interaction with the investigational products.

viii) Life expectancy < 1 year according to the judgment of the investigator.

ix) Active alcohol or substance use sufficient, in the investigator's opinion, to prevent adequate compliance with study therapy or to increase the risk of developing pancreatitis or chemical hepatitis.

x) History or ongoing psychiatry disorder.

xi) Any other clinical conditions or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for study or unable to comply with the dosing requirements.

- Physical and Laboratory Test Findings.

i) Screening laboratory analysis shows any of the following abnormal laboratory results:.

A. Grade IV glucose.

B. Grade IV electrolytes.

C. Grade IV transaminases.

D. Grade IV hematology.

ii) Calculated creatinine clearance < 60 mL/min as estimated by the Cockcroft-Gault equation.

* Allergies and Adverse Drug Reaction.

  i) Hypersensitivity to any component of the study drug formulations.
* Sex and Reproductive Status.

  i) Pregnancy.
* Other protocol-defined Inclusion/Exclusion criteria apply.

  i) Prisoners or subjects who are involuntarily incarcerated.

ii) Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2013-01-22 (Actual); Study Completion 2013-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 randomized and treated
Groups:
- Arm A: Reference Therapy: Atazanavir, heat-stable ritonavir [ATV/RTVHS] 300/100 mg QD + Tenofovir/emtricitabine [TDF/FTC] 300/200 mg QD by mouth for 48 weeks
- Arm B: Experimental Therapy: Atazanavir, heat-stable ritonavir [ATV/RTVHS] 300/100 mg QD + Lamivudine [3TC] 300 mg QD by mouth for 48 weeks
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Early termination of Study | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With HIV-1 RNA < 40 c/mL at Week 48
Description: Proportion of subjects with HIV-1 RNA < 40 c/mL at Week 48.
Time Frame: Week 48
Population: Week 48 not reached for any participant, data not collected at week 48
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Participants With HIV-1 RNA < 400 c/mL at Week 48
Description: Proportion of Participants with HIV-1 RNA < 400 c/mL at Week 48.
Time Frame: Week 48
Population: Week 48 not reached for any participant, data not collected at week 48
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion of Participants With HIV-1 RNA < 40 c/mL and < 400 c/mL at Week 96
Description: proportion of subjects with HIV-1 RNA < 40 c/mL and < 400 c/mL at Week 96.
Time Frame: Week 96
Population: Week 48 not reached for any participant, data not collected at week 96
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Adverse Events Through Weeks 48 and 96
Description: Incidence of Adverse Events through weeks 48 and 96 including serious adverse events (SAEs) and adverse events (AEs) leading to discontinuation.
  There were no SAEs or AEs reported in this early terminated study.
Time Frame: through weeks 48 and 96
Population: Week 48 and 96 not reached for any participant, data not collected through week 48 and 96
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Change From Baseline in eGFR and Bone Mineral Density at Weeks 48 and 96
Description: Percent change from baseline in eGFR and bone mineral density at weeks 48 and 96.
Time Frame: Weeks 48 and 96
Population: Week 48 and 96 not reached for any participant, data not collected at week 48 and 96
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Newly Emergent Genotypic Substitutions and Phenotypic Resistance to Study Drugs for Virologic Failures Through Week 48 and 96
Description: Incidence of newly emergent genotypic substitutions and phenotypic resistance to study drugs for virologic failures through Week 48 and 96.
Time Frame: Through week 48 and 96
Population: Week 48 and 96 not reached for any participant, data not collected through week 48 and 96
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: There were NO reported deaths among participants. There were NO adverse events or serious adverse events reported for any participant.
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.